CLINICAL TRIAL: NCT04771026
Title: The Effectiveness of Preemptive Nebulized Dexamethasone in Reducing Post- Operative Sore Throat Following the Use of AMBU® AURAGAINTM Device: A Double Blind, Randomised Clinical Trial
Brief Title: The Effectiveness of Preemptive Nebulized Dexamethasone in Reducing Post-Operative Sore Throat in Supraglottic Airway
Acronym: SGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Rhendra Hardy Mohamad Zaini, Associate Professor, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: USM/JEPeM/19120934
Record Dates: First submitted 2020-11-04; First posted 2021-02-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Sore Throat; Hoarseness; Dexamethasone; Supraglottic Airway Devices
Keywords: Dexamethasone; Supraglottic airway device; Post operative Sore throat; Post operative hoarseness of voice
MeSH Terms: conditions — Pharyngitis; Hoarseness | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Receiving routine conduct of general anaesthesia for supraglottic airway device
- Dexamethasone (Experimental): Receiving pre-operatively single dose nebulised dexamethasone 8mg prior to induction of general anaesthesia
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Pre-operatively nebuliser dexamethasone 8mg prior to induction of anesthesia
  Other Names: Decan
  Arms: Dexamethasone

SUMMARY:
This study aims to study the effectiveness of preoperatively nebulized dexamethasone in reducing the incidence and severity of Post Operative Sore Throat, POST in patients undergoing surgery under general anesthesia using the Ambu® AuraGainTM SGA device, with secondary aims of determining the effectiveness of dexamethasone in reducing post-operative cough severity and hoarseness of voice

DETAILED DESCRIPTION:
The role of dexamethasone in reducing the incidence and severity of postoperative sore throat (POST) with ETT use is established in few studies. Some of the studies had done were found to have result on pertaining to efficacy of steroids in reducing incidences of POST in usage of SGA device, hence we decided to undertake this double-blinded, randomized study in patients undergoing general anaesthesia using the Ambu® AuraGainTM SGA device.

Dexamethasone which is 26.6 and 6.6 more potent than cortisol and prednisolone, acts via anti-inflammatory effects; inhibiting and reducing the release of inflammatory mediators. Hence this study aims to study the effectiveness of preoperative nebulized dexamethasone in reducing the incidence and severity of POST to improve patient satisfaction following general anaesthesia,and reduce morbidity.

OBJECTIVES

General:

To determine the effectiveness of preoperatively nebulized dexamethasone in reducing the incidence of post-operative sore throat following Ambu® AuraGainTM SGA device use.

Specific:

1. To compare the incidence of post-operative sore throat (POST) with pre-operatively nebulized dexamethasone following insertion of Ambu® AuraGainTM SGA device at 30 minutes and 24 hours post operatively.
2. To compare the severity of POST with pre-operatively nebulized dexamethasone using a visual analogue scale (VAS) following insertion of Ambu® AuraGainTM SGA device at 30 minutes and 24 hours post-operatively.
3. To compare the incidence and severity of cough with pre-operatively nebulized dexamethasone using a 4-point scale grading at 30 minutes and 24 hours post-operatively following the insertion of Ambu® AuraGainTM SGA device.
4. To compare the incidence and severity of hoarseness of voice with pre-operatively nebulized dexamethasone using a 4-point scale grading at 30 minutes and 24 hours post-operatively following the insertion of Ambu® AuraGainTM SGA device.

HYPOTHESIS

Null hypothesis H0:

There is no difference in terms of efficacy of pre-operatively nebulised dexamethasone in reducing the incidence and severity of POST Sore throat, cough and hoarseness will be graded as per Tazeh-Kand et al's study

Alternative hypothesis H1:

Pre-operatively nebulised dexamethasone is effective in reducing the incidence and severity of POST Sore throat, cough and hoarseness will be graded as per Tazeh-Kand et al's study

RESEARCH DESIGN The proposed study design is a single-centre, randomized, double-blind, controlled, parallel-group interventional study conducted in Kelantan, Malaysia.

Patients will be randomized (using a block randomization software) to 2 study arms (1:1 ratio), into Groups C and D whereby:

Group C: Control group, patients receiving usual standard of care in practice of SGA device (including analgesics), without receiving any active drug.

Group D: Patients receiving nebulised dexamethasone 8mg (2ml) with 3mls of normal saline 0.9% 30 minutes prior to induction of anaesthesia in the pre-operative receiving room via a wall-mounted oxygen source at 15L/minute.

After randomization, each patient will stay in their assigned treatment arm for the duration of the study.

This will be a double-blinded randomized controlled study, carried out by a single operator and assessor. Both operator/ assessor and patient will be blinded.

STUDY AREA Operating theatres in Hospital Universiti Sains Malaysia, HUSM, Kubang Kerian.

INTERVENTIONS Group C: Control group, patients receiving usual standard of care in practice of SGA device (including analgesics), without receiving any active drug.

Group D: Patients receiving nebulised dexamethasone 8mg (2ml) with 3mls of normal saline 0.9% 30 minutes prior to induction of anaesthesia in the pre-operative receiving room via a wall-mounted oxygen source at 15L/minute.

SAMPLE SIZE ESTIMATION The sample size was estimated using the PS Software version 3.1.2 (Dupont and Plummer 1997) based on comparing 2 proportions for incidence of sore throat, And G*Power version 3.1.9.4 (Erdfelder, Faul, & Buchner, 1996) based on a 3 point scale for determining the severity of sore throat, cough and hoarseness of voice.

Where:

* Alpha: 0.05
* Power: 80%

Based on the parameters in the study by Tazeh-Kand NF, Eslami B, Mohammadian K. Inhaled fluticasone propionate reduces postoperative sore throat, cough, and hoarseness. Anesth Analg. 2010 Oct;111(4):895-8 (23).

The largest sample size generated was 128 (for 64 patients in each arm) for incidence of cough 1 hour post-operatively to detect a 30% difference in prevalence of cough between 2 study groups with a alpha value of 0.05 and power of 80%.

DATA COLLECTION METHOD After written consent pre-operatively, patients will be randomized as 2 groups

- Group C, and Group D. Group C: Patients receiving normal conduct of anaesthesia Group D: Patients receiving dexamethasone 8mg (2ml) with 3mls of normal saline 0.9%.

Patients will receive a sealed, opaque envelope containing a code with either N or D according to the randomization software pre-operatively, which will be opened by an anesthesiologist or nurse not involved in the study. The anesthesiologist or nurse opening the envelope will be told to withhold this information from the operator/investigator and patient. If the envelope contains the letter D, the said nurse/ anesthesiologist will be told to prepare and administer the nebulised drug as described, also without the knowledge of the operator/investigator. The operator/investigator will have no contact with the patient once the envelope is opened, and will remain away from the preoperative receiving room for 30 minutes from the arrival of patient.

Patients in group D will receive a total of 5mls of nebulized drug 30 minutes prior to induction of anaesthesia in the pre-operative receiving room via a wall-mounted oxygen source at 15L/minute.

After nebulisation for 30 minutes in the pre-operative receiving area, patients will be brought to the respective operating theatre. Monitoring according to standards will be applied - Non-invasive blood pressure, ECG, oxygen saturation, and capnography.

A humidified gas exchanger will be used for all patients.

Conduct of anesthesia will be as follows:

* Patients will not be premedicated
* Patients will be pre-oxygenated with 100% oxygen for 3-5 minutes or until an end-tidal oxygen fraction of 85 is achieved
* Intravenous induction with IV Fentanyl 1-2 mcg/kg, IV Propofol 1-3mg/kg, with no use of neuromuscular blockade of IV Dexamethasone.
* The insertion of a fully deflated SGA AMBU AURAGAIN® lubricated with Lignocaine 2% on the posterior aspect using the appropriate size according to patients' weight once there is loss of eyelash reflex by the operator using a standardized technique. The cuff will then be inflated with appropriate amount of air according to LMA size
* Cuff pressure will be measured immediately once the airway is secured, and subsequently measured hourly using a handheld pressure gauge. Cuff pressure of not more than 60 cmH20 will be maintained
* Anaesthesia will be maintained using Sevoflurane, titrated to a Minimum Alveolar Concentration (MAC) of 0.9-1.0 in 50/50 oxygen/air mixture with SIMV (Pressure or volume control) mode
* At the end of anaesthesia, the oral airway will be suctioned once gently and 100% oxygen will be administered until the SGA removed without deflation once regular, spontaneous ventilation has returned with opening of eyes to calling of name

Patients will be transferred to the recovery area where all patient will receive supplemental oxygen via face mask at 5L/minute until discharged from the post-operative recovery unit.

The 4 point questionnaire on POST will be applied at 30 minutes to 1 hour and 24 hours post-operatively in the ward by the same operator. If the patient is discharged prior to the 24 hour interview, they will be followed up via phone.

Scoring System for Sore Throat, Cough and Hoarseness, from Tazeh-kand et al:

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-70 years
* American Society of Anaesthesiology (ASA) physical status of 1 and 2
* Patients undergoing elective procedures under general anaesthesia between the data collection period suitable for SGA device

Exclusion Criteria:

* Pre-existing sore throat/hoarseness on pre-operative assessment
* Patients with history of postoperative nausea or vomiting
* Recent (2 weeks) upper or lower respiratory tract infection
* Known hypersensitivity to dexamethasone or on regular steroids
* Uncontrolled diabetes of capillary blood sugar more than 10mmol/l on pre-operative assessment
* Morbidly obese with BMI > 40 kg/m2
* Procedure exceeding 3 hours duration
* Procedure requiring prone or Trendelenburg position or manipulation of head post-induction
* Oral and neck surgeries
* Pregnant patients
* Patients with cognitive disabilities
* Patients requiring nasogastric tube or nasal temperature probe insertion
* Patient refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of POST up to 24 hours post-operatively in patients who received pre-operative nebulized dexamethasone | up to 24 hours post-operatively
  Patients will be evaluated using scoring system for sore throat, cough and hoarseness

SECONDARY OUTCOMES:
Incidence of cough up to 24 hours post-operatively in patients who received pre-operative nebulized dexamethasone | up to 24 hours post-operatively
  Patients will be evaluated using scoring system for sore throat, cough and hoarseness
Incidence of hoarseness of voice up to 24 hours post-operatively in patients who received pre-operative nebulized dexamethasone | up to 24 hours post-operatively
  Patients will be evaluated using scoring system for sore throat, cough and hoarseness

CONTACTS AND LOCATIONS:
Overall Officials: rhendra hardy Mohamad zaini, MD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- University of Science Malaysia Hospital, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No